CLINICAL TRIAL: NCT05813639
Title: EuroPainClinicsStudy XIr-Zj (Cryoablation vs Radiofrequency Ablation of Medial Nerve Branches of Dorsal Roots Crossing Z Joints)
Brief Title: EuroPainClinicsStudy XIr-Zj
Acronym: EPCS XIr-Zj
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Europainclinics z.ú. (Other)
Collaborators: Slovak Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6146/2022/ODDZ-25513
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Prospectively randomized patients with positive facet joint syndrome
Who Masked: Care Provider
Masking Description: sealed envelope, random software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbar medial branch cryoablation (Experimental): Lumbar medial branch cryoablation Procedure lumbar medial branch cryoablation Decreasing the electrode temperature to - 85 C for 120 seconds in two cycles. Follow-up: before the procedure, 3 months, 6 months, 12 months, and 24 months after the procedure Repeated cryoablation ablation procedures are allowed (when VAS will be =/> 4 ) Procedure/Surgery: Lumbar medial branch cryo ablation neurotomy A procedure based on positive lumbar Z- joint testing followed by medial branch neurotomy
  Interventions: Procedure: Lumbar medial branch cryo ablation neurotomy
- Lumbar medial branch RF neurotomy (Experimental): Lumbar medial branch RF neurotomy Procedure lumbar medial branch RF neurotomy: Raising the temperature of the tip of the electrode to 85 C for 120 seconds. RF generator. Follow-up: before the procedure, 3 months, 6 months, 12 months, and 24 months after the procedure. Repeated cryoablation ablation procedures are allowed (when VAS will be > 4 )
  Interventions: Procedure: Lumbar medial branch radiofrequency ablation neurotomy
- Lumbar fazet joint decapsulation (Experimental): Lumbar facet joint decapsulation through an endoscopic approach
  Interventions: Procedure: Endoscopic denervation of fazet joint

INTERVENTIONS:
Procedure: Lumbar medial branch cryo ablation neurotomy — The procedure is based on positive lumbar Z- joint testing followed by medial branch neurotomy
  Arms: Lumbar medial branch cryoablation
Procedure: Lumbar medial branch radiofrequency ablation neurotomy — The procedure is based on positive lumbar Z- joint testing followed by medial branch neurotomy
  Arms: Lumbar medial branch RF neurotomy
Procedure: Endoscopic denervation of fazet joint — The procedure is based on positive lumbar Z- joint testing followed by decapsulation of the facet joint through an endoscopic approach
  Arms: Lumbar fazet joint decapsulation

SUMMARY:
Determine the efficacy of lumbar medial branch neurotomy by radiofrequency and cryoablation in patients with chronic low back pain

DETAILED DESCRIPTION:
Facet joint pain encompasses a significant portion of the possible sources of pain in patients with vertebrogenic algic syndrome.A typical symptom caused by facet joint irritation of the medial branch nerve is a back pain with intermittent irregular patchy pain spreading to the legs. The cause of this pain is irritation of the medial branch of the dorsal nerve root which innervates a facet joint. Confirmation of the source of the pain involves local anaesthetic blocks of the medial nerve branches in several adjoining vertebral areas. If this test is positive, then the patient's condition is indicated for radiofrequency ablation or cryoablation of the nerve branches. Description of interventional procedures: Patients with chronic low back pain with confirmed zygapophysial joint pain after previous two medial branch nerve blocks with positive results are indicated for radiofrequency medial neurotomy or alternative cryoablation neurotomy. Navigation with probes in both cases is arranged and directed according to fluoroscopic imaging.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 20 and 80
* positive two medial branch nerve blocks with pain relief over 80% during the first 12 hours after nerve block application
* positive patient history of facet joint pain
* patients with chronic low back pain for at least 6 months with back pain and leg pain (VAS >=5)
* those who (only if a signature was obtainable), or whose legal guardian, fully understood the clinical trial details and signed the informed consent form

Exclusion Criteria:

* patients with a history of other spinal diseases (compression fracture, spondylitis, tumor)
* women with positive a pregnancy tests before the trial or who planned to become
* pregnant within the following 3 years
* other patients viewed as inappropriate by the staff
* disagreement with participation in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline EuroQoL-5 Dimension (EQ-5D) Value 6m | 6 months follow-up
  EQ-5D-5L self-care, usual activities, pain/discomfort and anxiety/depression
Change From Baseline EuroQoL-5 Dimension (EQ-5D) Value 12m | 12 months follow-up
  EQ-5D-5L self-care, usual activities, pain/discomfort and anxiety/depression
Change From Baseline Visual Analog Pain Scale (VAS) of Back Pain 6m | 6 months follow-up
  Change From Baseline Visual Analog Pain Scale (VAS) of Back Pain 6m measured by VAS 10 point measurement
Change From Baseline Visual Analog Pain Scale (VAS) of Back Pain 6m | 12 months follow-up
  Change From Baseline Visual Analog Pain Scale (VAS) of Back Pain 6m measured by VAS 10 point measurement
Oswestry Disability Index (ODI) 12m | 12 months follow-up
  The ODI self-administered questionnaire measuring 0-100 scale
Oswestry Disability Index (ODI) 6m | 6 months follow-up
  The ODI self-administered questionnaire measuring 0-100 scale

CONTACTS AND LOCATIONS:
Overall Officials: MD, PhD, FIPP Rapcan, MD, FIPP, Study Chair — R-Clinic Bardejov, Slovakia, 085 01
Locations (1):
- MD, PhD, FIPP Rapcan, Bardejov, Slovakia

IPD SHARING:
Plan to Share IPD: No
publishing results

REFERENCES:
- [Derived] Kocan L, Rapcan R, Mlaka J, Griger M, Poliak L, Lences P, Kovalicova L, Manik E, Sherdil N, Burianek M, Vaskova J. Comparative Effectiveness of Radiofrequency Ablation, Cryoablation, and Endoscopic Denervation for Lumbar Facet Pain: A Multicenter Trial. Spine (Phila Pa 1976). 2026 Jan 1;51(1):1-8. doi: 10.1097/BRS.0000000000005539. Epub 2025 Nov 4. PMID 41084911